CLINICAL TRIAL: NCT04067375
Title: Towards Routine HPA-screening in Pregnancy to Prevent FNAIT: Assessing Disease Burden and Optimising Risk Group Selection
Brief Title: Towards Routine HPA-screening In Pregnancy to Prevent FNAIT
Acronym: HIP
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Sanquin Research & Blood Bank Divisions (Other); Landsteiner Foundation for Blood Transfusion (Other)
Responsible Party: Principal Investigator, DickOepkes, Professor of Obstetrics and Fetal Therapy. Head of the section Fetal Medicine., Leiden University Medical Center
Other Study IDs: P16.002
Record Dates: First submitted 2019-07-16; First posted 2019-08-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Fetal and Neonatal Alloimmune Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Via a nationwide routine screening during pregnancy EDTA anticoagulated blood samples will be collected. Plasma and buffy coat will be stored.
  On plasma the following analysis will be performed:
  * HPA-1a typing by a new developed protol making use of ELISA.
  * Antibody screening by the Luminex assay.
  * Surface Plasmon Resonance on a sensor chip.
  To identify high risk cases fucosylation level of the antibodies will be performed. In addition to this the binding and functional effects to endothelial cells will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant women, HPA-1a positive: RhD or Rhc negative women, identified through prenatal screening for red cell alloimmunization, that are typed as HPA-1a positive.
  Interventions: Other: Clinical data collection.
- Pregnant women, HPA-1a negative with HPA-1a alloantibodies: RhD or Rhc negative women, identified through prenatal screening for red cell alloimmunization, that are typed as HPA-1a negative and have formed anti-HPA-1a alloantibodies.
  Interventions: Other: Clinical data collection.
- Pregnant women, HPA-1a negative without HPA-1a alloantibodies: RhD or Rhc negative women, identified through prenatal screening for red cell alloimmunization, that are typed as HPA-1a negative and did not have formed anti-HPA-1a alloantibodies.
  Interventions: Other: Clinical data collection.

INTERVENTIONS:
Other: Clinical data collection. — The following clinical data will be collected; maternal baseline characteristics, delivery related data, neonatal outcome, neonatal bleeding signs.

SUMMARY:
Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT) is the most common cause of severe thrombocytopenia in otherwise healthy born neonates. FNAIT results in a risk of bleeding the most severe complication being intracranial haemorraghes (ICH). Bleedings can be prevented by effective antental treatment. In the absence of screening programs this treatment is too late to prevent the first affected child. The investigators aim to identify the pregnancies at risk and describe the incidence and natural course of this disease. In this way fetuses at risk can be identified in the future and timely antenatal treatment can be initiated.

DETAILED DESCRIPTION:
Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT) is the most common cause of severe thrombocytopenia in neonates. It is an immunological process, in which Human Platelet Antigen (HPA) alloantibodies produced by the mother can cross the placenta and target fetal platelets. The most frequent alloantigen to elicit platelet-reactive antibody responses is HPA-1a. The resulting low platelet count in the fetus or neonate correlates with an increased risk of bleeding complications and severe adverse outcome, defined as perinatal death or intracranial haemorrhage (ICH). This can lead to life-long handicaps, cerebral palsy, cortical blindness and mental retardation. One in 50 pregnancies is at risk for FNAIT, since 2,1% of the Caucasian population is HPA-1a negative. Alloantibodies are calculated to be present in 1:400 pregnancies, leading to FNAIT-related severe adverse outcome in at least 1:1300 fetuses or neonates, and this is likely an underestimation. There is a highly effective antenatal treatment available for preventing these severe adverse outcomes, consisting of weekly injection of intravenous immunoglobulins (IvIG). Unfortunately, in the current practice, this treatment can only be applied in subsequent pregnancies with known alloimmunization, after a symptomatic sibling leading to diagnosis of the disease. In potential future antenatal screening for HPA-alloantibodies, all pregnancies at risk can be identified in time, to start antenatal treatment and reduce severe adverse outcomes. However, before such a program can be realised, detailed information about incidence and natural course of the disease is needed. Furthermore, laboratory tests to identify fetuses at high risk to prevent overtreatment are needed, since approximately 10-30% of the HPA alloimmunized cases result in severe thrombocytopenia and clinically relevant disease.

Objectives:

1. The main objective of this study is to assess the incidence and severity of FNAIT and bleeding complications (including ICH) among neonates.
2. To develop a screening platform, including diagnostic assay(s) to identify fetuses at high risk for bleeding complications due to FNAIT.

Study design: Prospective observational cohort

Study population: Pregnant women

Main study parameters/endpoints: The main study parameters are HPA-1a alloantibodies, clinically relevant FNAIT. Secondary parameters include: neonatal outcome (bleeding signs other than ICH, treatment for thrombocytopenia, morbidity).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: These pregnant women participate in the national antenatal screening programme for Prevention and Screening of Infectious diseases and Erythrocyte Immunisation (PSIE) and have a routine blood sampling at 27th week of gestation. This blood sample will be used this to perform all necessary tests, so no additional (medical) procedures will be performed. Additionally, after delivery clinical data concerning the pregnancy, delivery and the health of the child in the first postnatal period are collected by questioning the obstetric health care provider.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women, of whom routine blood samples are taken at 27 weeks gestational age (GA).

Exclusion Criteria:

* There are no predefined exclusion criteria, since we are aiming to determine the incidence in the complete pregnant population in the Netherlands.

[ WILSONBEKWAAM EXCLUSIE]

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 3660 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical relevant FNAIT | Within 7 days after birth.
  Incidence of HPA-1a mediated FNAIT. defined as severe or mild FNAIT
  Severe: Intracranial haemorrhage or Internal organ haemorrhage Mild: petechiae, hematoma, purpura or mucosal bleeding.Thrombocytopenia for platelet transfusion, IVIg or clinical observation.

SECONDARY OUTCOMES:
Neonatal thrombocytopenia | Within 7 days after birth.
  Thrombocytopenia: platelet count <150 x10^9/L Moderate thrombocytopenia: platelet count <100 x10^9/L Severe thrombocytopenia: platelet count <50 x10^9/L Extremely severe thrombocytopenia: platelet count <20 x10^9/L
Neonatal infection | Within 7 days after birth.
  CRP >10 and positive blood culture, for which antibiotics are administerd
Chromosomal abnormality | Within 7 days after birth.
  Chromosomal abnormalities as measured by DNA assessment (karyotyping, array, WGS/WES)

OTHER OUTCOMES:
Maternal age | Measured at 27 weeks gestational age of current pregnancy.
  Maternal age in years
Number of participatnts with idiopathic thrombocytopenic purpura | At inclusion
  Idiopathic thrombocytopenic purpura defined as thrombocytopenia in presence of autoantibodies.
Spontaneous miscarriage in obstetric history | At inclusion
  Number of previous spontaneous miscarriage before 12 weeks' gestation
Intrauterine fetal demise in obstetric history | At inclusion
  Number of previous IUFD after 12 weeks' gestation
Number of participants with hypertensive disorder | 3 months after delivery
  Pre-eclamspsia or pregnancy induced hypertension
Prematurity | through study completion, until delivery, an average of 6 months
  Gestational age at delivery below 37 weeks (premature) Or below 34 weeks gestation (very premature)
Apgar Score at 5 minutes after birth | 5 minutes after birth
  Measured as Apgar Score below 7 at 5 minutes after birth
Small for gestational age | through study completion, until delivery, an average of 6 months
  Birth weight (in grams) below the 10th percentile for the corresponding estational age at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dick Oepkes, Prof MD PhD, Study Director — Department of Obstetrics, Leiden University Medical Centre, Leiden; Masja de Haas, Prof MD PhD, Study Director — Department of Immunohematology Diagnostics, Sanquin Diagnostics, Amsterdam; Ellen vd Schoot, Prof MD PhD, Study Director — Department of Experimental Immunohematology, Sanquin Reseach, Amsterdam
Locations (1):
- Stichting Bloedbank Sanquin, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
No information will be given about individual participant data to the participating pregnant women, nor the obstetric caregiver will be informed about the serological HPA-1a typing results. Also, we decided to perform the antibody detection test after birth. Thus no additional information can be known that would otherwise change the management of the current pregnancy, according to the Dutch Guidelines.

REFERENCES:
- [Derived] de Vos TW, Winkelhorst D, Porcelijn L, Beaufort M, Oldert G, van der Bom JG, Lopriore E, Oepkes D, de Haas M, van der Schoot E. Natural history of human platelet antigen 1a-alloimmunised pregnancies: a prospective observational cohort study. Lancet Haematol. 2023 Dec;10(12):e985-e993. doi: 10.1016/S2352-3026(23)00271-5. Epub 2023 Oct 27. PMID 38407610
- [Derived] Winkelhorst D, de Vos TW, Kamphuis MM, Porcelijn L, Lopriore E, Oepkes D, van der Schoot CE, de Haas M. HIP (HPA-screening in pregnancy) study: protocol of a nationwide, prospective and observational study to assess incidence and natural history of fetal/neonatal alloimmune thrombocytopenia and identifying pregnancies at risk. BMJ Open. 2020 Jul 20;10(7):e034071. doi: 10.1136/bmjopen-2019-034071. PMID 32690731